CLINICAL TRIAL: NCT00750386
Title: Dose Dense Administration of Paclitaxel and Carboplatin Combination as 1st Line Treatment in Patients With Ovarian Carcinoma
Brief Title: Paclitaxel and Carboplatin Combination as 1st Line Treatment in Ovarian Carcinomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Christos Emmanouilides, Hellenic Oncology Research Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.07
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Ovarian Cancer
Keywords: Cancer; Ovarian cancer; Dose-dense chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Paclitaxel; Carboplatin

ARMS (1):
- 1 (Experimental): Paclitaxel/Carboplatin
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — 175 mg/m2, I.V, every 2 weeks
Drug: Carboplatin — Carboplatin AUC, I.V, 5 every 2 weeks

SUMMARY:
This trial will determine the feasibility and toxicity of dose intense (every 2 weeks) of paclitaxel+carboplatin combination following cytoreductive surgery in patients with stage Ic-IV ovarian cancer.

DETAILED DESCRIPTION:
Dose dense chemotherapy has been proven beneficial in various oncological settings. It is proposed that this concept be tested in ovarian cancer, with the support of growth factors. It is hypothesized that, if feasible, dose-dense chemotherapy may be more effective.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed ovarian cancer requiring standard chemotherapy
* Patients have to be chemotherapy naive
* Patients may have undergone cytoreductive surgery, or this may have been omitted due to dissemination
* Age >18 years.
* Performance status (WHO) 0-2
* Life expectancy of at least three months.
* Adequate bone marrow function (Absolute neutrophil count >1000/mm^3, Platelet count>100000/mm^3, Hemoglobin>9gr/mm^3).
* Adequate liver (Bilirubin<1.5 times upper limit of normal and SGOT/SGPT<2 times upper limit of normal) and renal function (creatinine<2mg/dl)
* Informed consent

Exclusion Criteria:

* Pregnant or nursing
* Psychiatric illness or social situation that would preclude study compliance'
* Other concurrent uncontrolled illness
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and the response rate | Toxicity assestment of the 1st cycle for the first 10 patients. Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment on each cycle
Time to tumor progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christos Emmanouilides, MD, Principal Investigator — Interbalkan Hospital, division of Oncology, Pylaia, Thessaloniki
Locations (12):
- Greece (12):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athnes, Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - Department of Medical Oncology, "Marika Iliadis" Hospital of Athens, Athens
  - Department of Medical Oncology, Air Forces Military Hospital of Athens, Athens
  - Medical Oncology Unit, 401 Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - First Department of Medical Oncology, "Metaxa's" Anticancer Hospital of Pireas, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki
  - Interbalkan Hospital, division of Oncology, Pylaia, Thessaloniki, Thessaloniki
  - Medical Oncology Unit, "AXEPA" General Hospital of Thessaloniki, Thessaloniki